CLINICAL TRIAL: NCT06817629
Title: Effects of Ventilation With Tidal Volume Adjusted on Driving Pressure on Ventilation/Perfusion Ratios and Hemodynamics in ARDS
Acronym: Hemodriving
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241429
Record Dates: First submitted 2025-01-07; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: ARDS
Keywords: ARDS; V/Q ratios; Hemodynamic
MeSH Terms: interventions — Hemodynamics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Effects of ventilation with tidal volume adjusted on driving pressure on ventilation/perfusion ratios and hemodynamics in ARDS — To ventilated patients with ARDS with an objective of driving pressure than a tidal volume set on predicted body weight

SUMMARY:
The driving pressure (DP) is defined as the pressure above the end-expiratory pressure (PEEP) required to distend the respiratory system by the tidal volume (Vt). It is calculated as follows: DP = Plateau pressure - PEEP. It is also equal to the ratio between the tidal volume and the compliance of the respiratory system (Crs): DP = Vt/Crs. Crs is correlated with end-expiratory lung volume, i.e., the lung volume available to receive the tidal volume. DP allows adaptation of the Vt to the available lung volume when the lungs are diseased, rather than to a fraction of lung size when they are healthy, as occurs when tidal volume is adjusted in mL/kg of predicted body weight (PBW). DP is therefore a better reflection of the deformation applied by the tidal volume and the risk of overdistension. It is an important prognostic indicator in acute respiratory distress syndrome (ARDS), with a risk of excess mortality when DP exceeds 14 cm H2O. Conversely, an excessively low DP, suggesting a low tidal volume in relation to the available lung volume, may theoretically also be accompanied by deleterious effects: de-recruitment, atelectrauma, the need to increase respiratory rate, the need for significant sedation, or even curarization. DP and Vt can influence hemodynamics, as overdistension is associated with an increase in dead space and the occurrence of acute cor pulmonale. On the other hand, de-recruitment due to low tidal volume can lead to hypoxic vasoconstriction with an increase in right ventricular afterload.

DETAILED DESCRIPTION:
It is hypothesized that ventilating ARDS patients with a tidal volume adjusted to mechanical power (MP) rather than 6 ml/kg of predicted body weight (PBW) is associated with improved ventilation/perfusion ratios and better right ventricular loading conditions. The objective is to evaluate the effects of ventilation with a tidal volume adjusted to target driving pressure (DP) between 12 and 14 cmH2O on ventilation/perfusion ratios in ARDS patients. The study consists of a standardization phase where patients receive ventilation with a tidal volume of 6 ml/kg PBW, with PEEP and FiO2 adjusted according to a PEEP/FiO2 table to maintain SpO2 between 90-95%. The respiratory rate will be clinician-adjusted, and settings will be maintained for 30 minutes. Following this, patients will undergo two randomized ventilation steps: (1) Vt-Vent, where settings remain identical to the standardization phase, and (2) DP-Vent, where tidal volume is adjusted to target a DP of 12-14 cmH2O while maintaining the same EtCO2 value as in the Vt-Vent phase. PEEP and FiO2 will remain unchanged. Data collection will begin at the 10th minute of each step.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ARDS moderate to severe according to the Berlin criteria
* Patient receiving continuous sedation and curarization
* Free and informed consent from the patient or family member

Exclusion Criteria:

* Pregnancy
* Adult patient subject to a legal protection measure (tutor, curator, etc.)
* Patients with a pacemaker, automatic implantable cardioverter defibrillator,
* Contraindications to thoracic belt placement (e.g., thoracic or spinal cord trauma, recent thoracic surgery)
* Undrained pneumothorax, bronchopleural fistula
* Hemodynamic instability (i.e., use of intravenous fluids of more than 10 mL/kg or vasopressors 2 mg/h of norepinephrine or 0.5 mg/h of epinephrine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with ARDS under deep sedation +/- paralized
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2027-03-05 (Estimated); Study Completion 2027-04-02 (Estimated)

PRIMARY OUTCOMES:
distribution of perfusion and ventilation across VA/Q ratios zones, wasted ventilation and perfusion. | 24 hours
  demonstration that ventilate patient with ARDS with an objective of protective driving pressure vent may change VA/Q ratio by using electrical impedance tomography

SECONDARY OUTCOMES:
DP-vent may induce a modification in patient with right ventricular | 24 hours
  RV/LV : right ventricle end-diastolic ratio
Change in right ventricular systolic function parameters | 24 hours
  Measurement of right ventricular systolic function measured in mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION